CLINICAL TRIAL: NCT00855491
Title: Prospective Evaluation of Posterior Capsule Opacification in Myopic Eyes 4 Years After AcrySof Single-Piece IOL Implantation
Brief Title: Posterior Capsule Opacification (PCO) With AcrySof Single-Piece IOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iladevi Cataract and IOL Research Center (Other)
Responsible Party: Dr. Shetal Raj, ICIRC
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 03-009
Record Dates: First submitted 2009-03-03; First posted 2009-03-04 (Estimated); Last update posted 2009-03-04 (Estimated); Status verified 2009-03

CONDITIONS: Posterior Capsule Opacification
Keywords: PCO; POCO

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1. MYOPIA (Experimental): axial length > 26.00 mm
  Interventions: Procedure: Phaco
- 2. Emmetropia (Active Comparator): emmetropic eyes- eyes with an axial length of 21.00 to 23.99 mm
  Interventions: Procedure: Phaco

INTERVENTIONS:
Procedure: Phaco — AcrySof Single-Piece IOL
  Other Names: emmetropic eyes; normal axial length

SUMMARY:
The purpose of this study what to evaluate if axial myopia might influence the development of PCO.

DETAILED DESCRIPTION:
We sought to prospectively compare PCO in eyes with myopia in relation to axial length with PCO in eyes with normal axial length, to decipher the role of axial myopia in PCO 4 years after surgery for senile cataract.

ELIGIBILITY:
Inclusion Criteria:

* local residency and presence of a cataract in an otherwise normal eye.
* Patients older than 50 years
* a dilated pupil after mydriasis
* Patients with retinochoroidal atrophy, retinal laser prophylaxis,
* hypertension

Exclusion Criteria:

* nondilating pupil after maximal dilation;
* pseudoexfoliation; mature, traumatic, black, or complicated cataracts;
* previous intraocular surgery;
* previous surgery for glaucoma;
* uveitis
* diabetes mellitus
* Patients who did not give consent preoperatively

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2003-07; Primary Completion 2004-09 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
the percentage area of PCO with posterior capsule opacity (POCO) software | 4 years

SECONDARY OUTCOMES:
the presence of PCO within the central 3-mm zone were noted | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: ALPESH SHAH, MS, Principal Investigator — Iladevi Cataract and IOL Research Center
Locations (1):
- Raghudeep Eye Clinic, Ahmedabad, Gujarat, India